CLINICAL TRIAL: NCT03872466
Title: Glove Rehabilitation Application for Stroke Patients (GRASP)
Brief Title: Glove Rehabilitation Application for Stroke Patients
Acronym: GRASP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barron Associates, Inc. (Industry)
Collaborators: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GRASP
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Occupational Therapy; Virtual Reality

STUDY DESIGN:
Intervention Model Description: Intervention group performs therapy using the GRASP system for virtual world-based practice.
  Control group follows a Usual Care Treatment (UCT) regimen.
Who Masked: Investigator
Masking Description: Investigator administrating assessments will be blinded to subject group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- GRASP Intervention (Experimental): This arm will perform eight weeks of independent home practice for upper extremity therapy using the GRASP system.
  Interventions: Device: GRASP HEP
- Control (Active Comparator): Participants in the control group will continue to receive any previously prescribed therapy services. These patients will not receive any treatment services through the study as control group participants.
  Interventions: Behavioral: Usual Care Treatment (UCT)

INTERVENTIONS:
Device: GRASP HEP — The GRASP system comprises a sensor package and therapy game software that works with a commercial glove orthosis to enable virtual world-based practice of activities of daily living (ADLs) involving the hand.
  Arms: GRASP Intervention
Behavioral: Usual Care Treatment (UCT) — Participants in the control group will continue to receive any previously prescribed therapy services. These patients will not receive any treatment services through the study as UCT group participants.
  Arms: Control

SUMMARY:
The University of Virginia (UVA) Director of Neurorehabilitation will lead GRASP randomized, controlled efficacy trials. The study will involve employment of the GRASP system in three one-hour sessions per week over eight weeks by stroke survivors suffering from ongoing hand function impairment.

DETAILED DESCRIPTION:
Testing will involve employment of the GRASP system (glove orthosis, sensor package, and application software) in three one-hour sessions per week over eight weeks by stroke survivors suffering from ongoing hand function impairment. This frequency and duration is consistent with previous studies successfully investigating new upper extremity (UE) therapies. The primary outcome of the efficacy study will be change in hand function for a group of participants using the GRASP system versus a control group receiving standard care over the same period.

Participants assigned to the GRASP intervention group will attend five outpatient clinic visits for consent, pre-assessment, and familiarization with the system, followed by an initial home visit and eight weeks (3x per week) of independent at-home practice. In this study period, GRASP intervention group participants will employ the instrumented glove orthosis while performing functional tasks within virtual activities of daily living (ADLs).

Participants in the Usual Care Treatment (UCT) control group will continue to receive any previously prescribed therapy services. These patients will not receive any treatment services through the study as UCT control group participants.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has had a right or left hemispheric stroke affecting normal hand function;
2. Participant has sufficient active finger flexion at the MCP joint in at least one finger to be detected by visual observation by a study therapist;
3. Participant has visual acuity with corrective lenses of 20/50 or better;
4. Participant's affected hand fits within sizing available for the glove orthosis;
5. Participant is no longer in an active UE rehabilitation program; and
6. Participant is currently living at a private residence and anticipates remaining at that location for the duration of study participation.

Exclusion Criteria:

1. Withholding or withdrawal of consent by the participant;
2. Inability to understand and follow verbal directions;
3. Determination by the Principal Investigator that participation would result in overexertion or significant discomfort or pain;

(3) A psychological diagnosis that in the determination of the Principal Investigator could significantly impact subject's participation or that could be aggravated by study participation (Principal Investigator will consult with candidate's personal physician as appropriate); (4) Determination by the Principal Investigator that participation would result in significant agitation or elevated stress; (5) Visual field deficit in either eye that impairs the ability to view the computer monitor; (6) Stiffness or contractures of the muscles, joints, tendons, ligaments, or skin that restricts normal movement; (7) More than mild tone/spasticity (measured on modified Ashworth, 5-point scale); (8) Severe contractures or joint deformities in the fingers; (9) Open wound or infection, severe edema, or excessive swelling which might interfere with wearing the glove; (10) Severe pre-stroke co-morbidities, such as cardiovascular, neurological, orthopedic, or rheumatoid impairments before stroke that may interfere with task performance; (11) Severe sensory deficits from the involved UE; or (12) Hemispatial neglect that impairs the ability to process and perceive visual stimuli provided through the computer monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UVA Outpatient Rehabilitation Clinic, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adams RJ, Ellington AL, Kuccera KA, Leaman H, Smithson C, Patrie JT. Telehealth-Guided Virtual Reality for Recovery of Upper Extremity Function Following Stroke. OTJR (Thorofare N J). 2023 Jul;43(3):446-456. doi: 10.1177/15394492231158375. Epub 2023 Mar 24. PMID 36960762

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GRASP Intervention | Control
Started | 12 | 9
Completed | 9 | 9
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GRASP Intervention | Control | Total
Number analyzed (Participants) | 12 | 9 | 21
Age, Continuous [Median (Full Range); unit: years] | 62 [45 to 82] | 60 [34 to 86] | 60 [34 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 9 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 9 | 8 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Pre Intervention Fugl-Meyer Assessment of Upper Extremity Motor Function (FMUE)
Description: FMUE is one of the most widely used and accepted quantitative measures of motor function in stroke patients, used in clinical and research settings. Individual patient movements associated with specific motor functions are scored using a 3-point ordinal scale (0, 1, or 2). The study employs a subscale of the full assessment that incorporates 33 items relevant to shoulder, elbow, forearm, wrist, hand, and grasp function, thus creating a possible range of 0 to 66 points. Higher scores correspond to higher levels of motor function.
Time Frame: Pre-intervention at Baseline
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | GRASP Intervention | Control
Number analyzed (Participants) | 9 | 9
score on a scale | 42.22 [35.66 to 48.78] | 42.44 [35.89 to 49.00]

2. Primary Outcome: Post Intervention Fugl-Meyer Assessment of Upper Extremity Motor Function (FMUE)
Description: as for outcome 1
Time Frame: Post Intervention at 8 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | GRASP Intervention | Control
Number analyzed (Participants) | 9 | 9
score on a scale | 52.33 [45.77 to 58.89] | 44.00 [37.44 to 50.56]

3. Secondary Outcome: Pre Intervention Wolf Motor Function Test Functional Assessment (WMFT-FA)
Description: The WMFT test is a functionally-oriented clinical and research instrument. The test consists of 15 motor tasks scored both for time and quality of movement.
  The WMFT Functional Assessment (WMFT-FA) score is an observational assessment of movement quality and scored using a 6-point ordinal rating scale that ranges from 0 (no use of the affected side attempted) to 5 (normal function). A total WMFT-FA score is calculated by taking the average across all 15 UE tasks. A patient's WMFT-FA score is thus a real number that can range from 0 to 5. An increase in WMFT-FA score implies improved motor function.
Time Frame: Pre-intervention at Baseline
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | GRASP Intervention | Control
Number analyzed (Participants) | 9 | 9
score on a scale | 2.70 [2.20 to 3.19] | 2.67 [2.17 to 3.16]

4. Secondary Outcome: Post Intervention Wolf Motor Function Test Functional Assessment (WMFT-FA)
Description: as for outcome 3
Time Frame: Post Intervention at 8 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | GRASP Intervention | Control
Number analyzed (Participants) | 9 | 9
score on a scale | 3.42 [2.73 to 4.12] | 2.84 [2.14 to 3.53]

5. Secondary Outcome: Pre Intervention Wolf Motor Function Test Time (WMFT-TIME)
Description: The WMFT test is a functionally-oriented clinical and research instrument. The test consists of 15 motor tasks scored both for time and quality of movement. WMFT-TIME is a quantitative measure calculated using the average time to complete the tasks. Any time greater than 120 seconds is recorded as 120 seconds. A patient's WMFT-TIME score (average completion time) thus ranges from 0 to 120. A reduction in WMFT-TIME implies improved motor function.
Time Frame: Pre-intervention at Baseline
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | GRASP Intervention | Control
Number analyzed (Participants) | 9 | 9
score on a scale | 8.52 [4.49 to 16.17] | 11.01 [5.80 to 20.90]

6. Secondary Outcome: Post Intervention Wolf Motor Function Test Time (WMFT-TIME)
Description: as for outcome 5
Time Frame: Post Intervention at 8 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | GRASP Intervention | Control
Number analyzed (Participants) | 9 | 9
score on a scale | 6.97 [3.67 to 13.24] | 7.46 [3.93 to 14.16]

7. Secondary Outcome: Pre Intervention Box and Blocks Test (BBT)
Description: The BBT provides a measure of unilateral gross manual dexterity. Subjects are asked to move 2.5 cm wooden cubes from one 8.5 cm tall box to another, as quickly as possible. The BBT score is simply the number of blocks moved in 60 seconds. A patient's WMFT-FA score is thus an integer number if blocks that is greater than or equal to zero. The maximum number of blocks is 150. An increase in BBT score implies improved motor function.
Time Frame: Pre-intervention at Baseline
Measure: Mean (95% Confidence Interval); unit: blocks
Arm/Group | GRASP Intervention | Control
Number analyzed (Participants) | 9 | 9
blocks | 22.89 [15.29 to 34.26] | 12.78 [6.48 to 25.19]

8. Secondary Outcome: Post Intervention Box and Blocks Test (BBT)
Description: as for outcome 7
Time Frame: Post Intervention at 8 weeks
Measure: Mean (95% Confidence Interval); unit: blocks
Arm/Group | GRASP Intervention | Control
Number analyzed (Participants) | 9 | 9
blocks | 28.44 [20.85 to 38.81] | 14.44 [7.76 to 26.88]

9. Secondary Outcome: Pre Intervention Motor Activity Log - Amount (MAL-Amount)
Description: The MAL is a structured interview assessing use of the affected arm in 30 daily activities in the subject's real-life experience. These range from turning on a light to eating finger foods. For each activity, the subject provides a self-assessment of the frequency with which the affected arm is involved in the activity (MAL-Amount) and the quality with which the affected arm performs (MAL-How Well). Grading is on a Likert scale. At the low end, 0 corresponds to never using the weaker arm for the activity. On the upper end, 5 corresponds to using the weaker arm equivalently to the stronger arm. A total MAL-Amount score is calculated by taking the average across all 30 activities. Likewise, a total MAL-How Well score is calculated by taking the average across all 30 activities. A patient's MAL-Amount and MAL-How Well scores are thus real numbers that can range from 0 to 5. An increase in these scores implies improved motor function.
Time Frame: Pre-intervention at Baseline
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | GRASP Intervention | Control
Number analyzed (Participants) | 9 | 9
score on a scale | 1.33 [0.80 to 1.86] | 1.30 [0.77 to 1.83]

10. Secondary Outcome: Post Intervention Motor Activity Log - Amount (MAL-Amount)
Description: as for outcome 9
Time Frame: Post Intervention at 8 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | GRASP Intervention | Control
Number analyzed (Participants) | 9 | 9
score on a scale | 2.55 [1.84 to 3.25] | 1.18 [0.48 to 1.89]

11. Secondary Outcome: Pre Intervention Motor Activity Log - How Well (MAL-How Well)
Description: as for outcome 9
Time Frame: Pre-intervention at Baseline
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | GRASP Intervention | Control
Number analyzed (Participants) | 9 | 9
score on a scale | 1.35 [0.79 to 1.91] | 1.18 [0.62 to 1.74]

12. Secondary Outcome: Post Intervention Motor Activity Log - How Well (MAL-How Well)
Description: as for outcome 9
Time Frame: Post Intervention at 8 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | GRASP Intervention | Control
Number analyzed (Participants) | 9 | 9
score on a scale | 2.70 [2.06 to 3.34] | 1.20 [0.56 to 1.84]

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | GRASP Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 0/12 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT03872466/Prot_SAP_000.pdf